CLINICAL TRIAL: NCT04403282
Title: Topical Eflornithine Hydrochloride for Pseudofolliculitis Barbae: A Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: Topical Eflornithine for Pseudofolliculitis Barbae: Randomized Controlled Trial
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Vaniqa no longer manufactured
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WRNMMC-2020-0298
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Pseudofolliculitis Barbae
Keywords: Pseudofolliculitis Barbae; Eflornithine
MeSH Terms: conditions — pseudofolliculitis barbae | interventions — Eflornithine

STUDY DESIGN:
Intervention Model Description: randomized, double-blinded, placebo-controlled, paired (right and left neck) comparison study examining eflornithine versus placebo for the treatment of PFB.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Paired(right and left neck) comparison group eflornithine (Active Comparator): randomized, double-blinded, placebo-controlled, paired (right and left neck) comparison study examining eflornithine versus placebo for the treatment of PFB.
  Interventions: Drug: Eflornithine Topical
- Paired(right and left neck) comparison group placebo (Placebo Comparator): randomized, double-blinded, placebo-controlled, paired (right and left neck) comparison study examining eflornithine versus placebo for the treatment of PFB.
  Interventions: Drug: Placebo Eflornithine Topical

INTERVENTIONS:
Drug: Eflornithine Topical — Subjects will apply placebo to one side of beard and eflornithine to other side for 16 weeks.
  Arms: Paired(right and left neck) comparison group eflornithine
Drug: Placebo Eflornithine Topical — Subjects will apply placebo to one side of beard and eflornithine to other side for 16 weeks.
  Arms: Paired(right and left neck) comparison group placebo

SUMMARY:
To study the efficacy of topical eflornithine for pseudofolliculitis barbae from a quality of life standpoint and with objective physician-measured lesion counts. Our hypothesis is that the hair growth retardation that occurs with eflornithine will perhaps reduce the frequency over time that service members need to shave which could improve the formation of PFB lesions.

DETAILED DESCRIPTION:
Pseudofolliculitis barbae (PFB), or 'ingrown hairs,' is a common skin disease of the face and neck caused by shaving in predisposed individuals who have naturally curly hair. It affects a disproportionate number of African American Service Members - up to 45% in one study.(Alexander, 1974) Keeping a close shave is a requirement for service in all of the Unites States armed services, and as a result, PFB is a major cause of morbidity in this population. The main rationale behind this policy is that a beard prevents a proper seal when using breathing protection devices, in particular gas masks. A review of various dermatologic conditions seen in wartime found that the incidence of PFB was 5.9% during the Vietnam War and 1.8% during Operation Iraqi Freedom (OIF) (Gelman, 2015). The authors argued that this was due to a relaxing of the shaving standards as part of the update PFB protocol followed during OIF. However, the United States Navy recently announced a change to their PFB protocol, discontinuing the issuance of permanent "no-shave" chits. Laser hair removal (LHR) using the Neodymium: Yttrium-Garnet (Nd:Yag) laser is the current treatment of choice for the majority of patients who fail conservative treatment with topical retinoids, antibiotics, and optimization of shaving practices. However, LHR treatment can induce a permanent change in facial hair density and patients treated with this modality may have to accept a permanent change in their ability to grow a beard. In addition, laser treatments have a potential for operative discomfort along with blistering and dyspigmentation of skin. Eflornithine is a topical medication that is FDA indicated for the treatment of unwanted terminal hairs in women. It works by its action as an irreversible inhibitor of ornithine decarboxylase, an enzyme responsible for the formation of polyamines which allow for various proliferative activities in the skin. It is the only known topical treatment that can retard the growth of human hair. Xia et al. showed that this medication can be used in conjunction with LHR to enhance the efficacy of the treatment for PFB(Xia, 2012). However, there are no studies to date that look at eflornithine as monotherapy for the treatment of PFB. The Unites States Navy has included topical eflornithine as a potential PFB treatment in their latest Bureau of Medicine and Surgery (BUMED) instruction despite the lack of evidence behind its use. If shown to be efficacious, this medication would provide a cost-effective treatment for PFB, especially in medical practices that do not have a hair removal laser. In addition, the effects of eflornithine are reversible with discontinuation, making it an ideal choice for patients and service members who would like to retain their ability to grow normal beards.

Goal: To study the efficacy of topical eflornithine for pseudofolliculitis barbae from an objective physician-measured lesion count. Our hypothesis is that the hair growth retardation that occurs with eflornithine will perhaps reduce the frequency over time that service members need to shave which could improve the formation of PFB lesions.

Plan

1. Recruitment of patients that meet inclusion criteria (No LHR treatments in the past year, Not pregnant or breast feeding).
2. Provide written informed consent.
3. Patients instructed to discontinue all other treatment modalities for PFB (plucking, waxing, chemical depilatories, topical retinoids).
4. Patients receive two identical 30-g jars from the Walter Reed Army Medical Center research pharmacist. The jars will be labeled "left" and "right" and randomized by the pharmacy using a random number generator.
5. Initial lesion counts and Skin Disease on Quality of Life survey measurements taken. Two (left and right) 2-cm circles drawn at the junction of the submental chin and anterior neck for the lesion counts.
6. Patients begin applying a thin layer of each cream corresponding to the site of application (left and right beard) twice a day.
7. Follow up at 4 week intervals, at which the number of hairs and inflammatory papules will be counted within the two 2-cm circles on the submental chin by two dermatology residents or staff dermatologists.
8. Patient then goes to research pharmacist. Pharmacist weighs both eflornithine as well as placebo cream to measure compliance. Re-issue new 30-g jars.
9. At week 16, final lesions counts administered.
10. Data is analyzed using Wilcoxon signed-rank tests.
11. Findings published.

ELIGIBILITY:
Inclusion Criteria:

* Active Duty Service Members with Pseudofolliculitis Barbae

Exclusion Criteria:

* Previous treatment with laser hair removal in the previous 12 months, Currently pregnant, seeking pregnancy, or breast feeding

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2020-09-27 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
number of skin lesions | 16 weeks
  number of skin lesions

SECONDARY OUTCOMES:
number of hairs | 16 weeks
  number of hairs

CONTACTS AND LOCATIONS:
Overall Officials: Sunghun Cho, MD, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
The PI will compile the names of the patients who are followed through week 16 in order to create the master subject list. Using the information stored on the master subject list (name, social security number, Medical Record Number), the research team will obtain data electronically from the patient medical records. Specifically, the lesion and hair counts on the face will be acquired. This will be recorded on the master data sheet. The master subject list will be password protected and only accessible to study personnel within the Walter Reed National Military Medical Center (WRNMMC) network. The master data sheet will be coded and available to the investigators and may be shared with research assistants or statisticians.

REFERENCES:
- [Background] Alexander AM, Delph WI. Pseudofolliculitis barbae in the military. A medical, administrative and social problem. J Natl Med Assoc. 1974 Nov;66(6):459-64, 479. No abstract available. PMID 4436875
- [Background] Gelman AB, Norton SA, Valdes-Rodriguez R, Yosipovitch G. A review of skin conditions in modern warfare and peacekeeping operations. Mil Med. 2015 Jan;180(1):32-7. doi: 10.7205/MILMED-D-14-00240. PMID 25562855
- [Background] Ogunbiyi A. Pseudofolliculitis barbae; current treatment options. Clin Cosmet Investig Dermatol. 2019 Apr 16;12:241-247. doi: 10.2147/CCID.S149250. eCollection 2019. PMID 31354326
- [Background] Xia Y, Cho S, Howard RS, Maggio KL. Topical eflornithine hydrochloride improves the effectiveness of standard laser hair removal for treating pseudofolliculitis barbae: a randomized, double-blinded, placebo-controlled trial. J Am Acad Dermatol. 2012 Oct;67(4):694-9. doi: 10.1016/j.jaad.2011.10.029. Epub 2012 Jan 9. PMID 22226431